CLINICAL TRIAL: NCT01788202
Title: An Observational, Prospective Study in Patients With Positive Urine Cocaine Metabolites Undergoing Surgery for General Anesthesia
Brief Title: Patients With Positive Urine Cocaine Metabolites Undergoing General Anesthesia
Status: Terminated | Type: Observational
Why Stopped: unable to enroll patients
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 0120090260
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Emergent Surgery
Keywords: cocaine and general anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
When it is safe to administer general anesthesia to the patient with cocaine positive urine drug screen has never been clearly determined. The study doctors would like to determine the effect of cocaine on blood pressure, heart rate and rhythm during surgery. After surgery, the subjects will be observed in regards to mental status and any changes in heart rate and rhythm.

DETAILED DESCRIPTION:
The risks associated with administering general anesthesia to cocaine abusing patients with a positive urine cocaine metabolite is a major cause of cancellation of surgery in many trauma centers. Although many clinicians wait 24 to 48 hours after a positive urine drug screen before administering anesthesia, no standard or practical guidelines have yet to determine when it is safe to proceed with general anesthesia in this patient population. Due to the lack of guidelines for these cases, the rate of cancellation of procedures for these patients is high. The frequent cancelling of such cases causes a waste of resources, personnel, and time. The risks associated with cocaine use that cause most clinicians to cancel cases are mainly due to the cardiovascular effects of cocaine. Increases in blood pressure, heart rate, temperature, and the potential for myocardial infarction and fatal arrhythmias are what clinicians fear when administering general anesthesia to these patients. However, due to the urgency of some of the cases, it would be beneficial to both the patient and institutions to know when it is safe to proceed with the case and when it is not. When it is safe to administer general anesthesia to the patient with cocaine positive urine drug screen has never been clearly determined. This observational study will evaluate the effects of general anesthesia on the cocaine abusing patient with cocaine positive urine drug screen.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists rating of 1-111
* Positive cocaine metabolite
* urgent surgery for acute abdomen, orthopedic trauma, maxillary-facial trauma

Exclusion Criteria:

* Failure to provide consent
* females who are pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects requiring urgent surgeries for acute abdomen, orthopedic trauma and maxillary facial trauma cases.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
cardiac arrythmia | intraoperatively
  Did the patient require rescue medication for cardiac arrythmia such as tachycardia or ST segment elevation on EKG strip

SECONDARY OUTCOMES:
hypotension | intraoperatively
  did subject require rescue for intraoperative hypotension

OTHER OUTCOMES:
Neurological deficit | post operatively to 24 hours
  does the subject display post operatively neurological def

CONTACTS AND LOCATIONS:
Overall Officials: J. Daniel Eloy, MD, Principal Investigator — UMDNJ/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No